CLINICAL TRIAL: NCT03681028
Title: Pilot Study Testing Feasibility of Individualized Therapy for Recurrent Glioblastoma
Brief Title: Feasibility of Individualized Therapy for Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer Clarke (Other)
Responsible Party: Sponsor-Investigator, Jennifer Clarke, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18108; NCI-2018-02194 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Glioblastoma
Keywords: Glioblastoma; Adult Glioblastoma; Glioma; Precision Medicine; Specialized Tumor Board
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Individualized therapy (Other): Study treatment for a given patient will consist of a regimen chosen from agents implicated in critical molecular signaling pathways and/or from signature-based predictions of drug efficacy. All agents are listed in the current pharmacopoeia for human use, but will differ amongst individual subjects. The study treatment will consist of up to 4 FDA approved drugs that have known dosing. This study is not only looking at 4 drugs. It is selecting up to 4 drugs per patient but the drugs chosen can be any FDA-approved drug. Therefore, it is not possible to pre-specify the medications.
  Interventions: Drug: Individualized therapy

INTERVENTIONS:
Drug: Individualized therapy — 1. For a given proposed individualized combination of drugs the first priority to establish doses will be to identify the same combination of drugs in a peer-reviewed journal article or presented as a reviewed abstract.
  2. When a proposed individualized combination of drugs has not previously been reported, the process to establish doses will be to then identify individual members of the proposed combination that have been used in combination with other cytotoxic agents similar to those being considered for combination therapy.
  3. When a proposed individualized combination of drugs has no available combination data, dosing guidelines will start with the FDA-approved package insert recommended dose.

SUMMARY:
The current study will test the ability and likelihood of successfully implementing individualized combination treatment recommendations for adult patients with surgically-resectable recurrent glioblastoma in a timely fashion. Collected tumor tissue and blood will be examined using a new diagnostic testing called University of California, San Francisco (UCSF) 500 Cancer Gene Panel which is done at the UCSF Clinical Cancer Genomics Laboratory. The UCSF 500 Cancer Gene Panel will help identify genetic changes in the DNA of a patient's cancer, which helps oncologists improve treatment by identifying targeted therapies.

DETAILED DESCRIPTION:
This is a single arm, non-randomized open-label study to assess feasibility of implementing an individualized treatment regimen in patients with surgical recurrent glioblastoma (GBM). Patients are not stratified according to demographic or treatment-related parameters. Patients must have recurrent glioblastoma treated with appropriate tumor treatment including radiation therapy at initial diagnosis. Surgery must be clinically indicated and patients must be candidates for tumor resection at UCSF.

The goal of the current study is to build upon prior results by confirming the feasibility of actually implementing patient-specific drug regimens in a rapid, clinically-relevant timetable. The investigators will also assess for efficacy, safety, and response outcomes of these patient-specific regimens, to generate preliminary data that would support a larger trial assessing efficacy of such an approach.

Resected tumor tissue and blood will be examined using Next Generation Sequencing (NGS) UCSF 500 Cancer Gene Panel at the UCSF Clinical Cancer Genomics Laboratory and Whole genome and RNA sequencing. The clinical report generated from the NGS UCSF 500 panel will be provided to a study-specific Tumor Board who will generate an individualized treatment recommendation based on the report. The individualized treatment regimen potentially will include up to 4 re-purposed, off-the-shelf, FDA-approved targeted agents. The Board will identify the expected/anticipated drug-drug interactions and anticipated additional toxicities of the combination of therapies. The treating physician is given the report, discusses the suggested treatment options with the patient, and initiates treatment, ideally within 28 calendar days (and no later than 35 calendar days) after surgery.

Patients may continue treatment until tumor progression, intolerable side effects, or patient/physician choice to discontinue.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age must be >= 18 years
2. Patients must understand and provide written informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization authorization prior to initiation of any study-specific procedures
3. Patients must have recurrence of histologically-proven glioblastoma or gliosarcoma, World Health Organization (WHO) grade IV that is surgically resectable.
4. The patient's surgeon thinks that they can resect at least 500 mg of tumor.
5. Patient must have Karnofsky Performance Scale (KPS) score >=70
6. Patient must have an estimated life expectancy ≥ 3 months
7. Patients may enroll independent of number of prior therapies or cumulative doses of prior therapies, but must have received appropriate prior therapy for GBM at time of initial diagnosis, including radiation therapy.
8. Patient must have adequate bone marrow function, renal function, and hepatic function as defined below:

   Adequate bone marrow function:
   1. absolute neutrophil count (ANC) >= 1,500/μL
   2. Platelets >= 100,000/μL

   Adequate hepatic function:
   1. total bilirubin <= 1.5x institutional upper limit of normal
   2. Aspartate aminotransferase (AST) /serum glutamic-oxaloacetic transaminase (SGOT) <= 2.5x institutional upper limit of normal
   3. Alanine aminotransferase (ALT) / serum glutamic-pyruvic transaminase (SGPT) <= 2.5x institutional upper limit of normal

   Adequate renal function:

   a. creatinine <= 1.5x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m2
9. Must be able to undergo MRI scans for tumor evaluation.
10. Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days prior to surgery.

    The effects of study drugs, either individually or their combination on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation and for 3 months after completion of study drug administration. The use of adequate contraception may be longer than 3 months depending on the drugs used and the FDA-approved labeling in cases of recommendation for contraception. Adequate contraception may include hormonal contraception, barrier method (condom, contraceptive sponge, diaphragm or ring), intrauterine device (IUD), tubal ligation, vasectomy and abstinence. Should a woman become pregnant (or suspect that she is pregnant) while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of study drug administration. Patient must not be a woman who is currently pregnant, due to the potential for teratogenic or abortifacient effects of study drugs, either alone or in combination. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with study drugs, lactating women who are breastfeeding should discontinue breastfeeding if the mother is treated with any study drug.
11. Patients must not have New York Heart Association (NYHA) Grade II or greater congestive heart failure
12. Patients must not have history of myocardial infarction or unstable angina within 12 months prior to study enrollment.

Exclusion Criteria:

1. Patient who has been treated with any chemotherapy or radiotherapy ≤4 weeks prior to date of study registration. Exceptions to this include: must be ≥ 23 days from last dose of temozolomide (TMZ), must be ≥ 6 weeks from last dose of nitrosurea.
2. Patient who has not recovered to grade 1 or baseline from the adverse effects of prior radiotherapy or chemotherapy.
3. Patient who is < 12 weeks from initial course of radiation
4. Patients with multifocal tumor, primarily infratentorial or posterior fossa tumor, or leptomeningeal dissemination of tumor.
5. Patient with any other active malignancy besides GBM, excluding non-melanomatous skin cancer, or carcinoma in situ of the cervix, prostate, or breast, unless patient has been disease-free/in remission for >=2 years prior to date of study enrollment
6. Patients known to be HIV-positive. HIV testing is not required for study participation.
7. Uncontrolled concurrent illness including psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent.
8. Any other acute or chronic medical or psychiatric condition, or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results, and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have successfully initiated therapy | Up to 35 days after surgery
  Feasibility of implementing a truly personalized tumor treatment drug regimen for patients with surgically resectable recurrent glioblastoma is defined as the percentage of patients who have successfully initiated therapy based on their individualized treatment regimen within 35 days following surgical resection of recurrent tumor.
Overall survival at 9 months (OS) | Up to 9 months
  Overall survival is defined as the length of time from start of individual treatment or combination treatment regimen until 270 days, or 9 months. For the participants who were alive at the end of study or lost to follow-up, overall survival will be censored on the last date when participants were known to be alive. OS will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Incidence of treatment-related Adverse Events (AEs) | Up to 1 year
  Incidence of treatment-related AEs, grades 3-5 using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 either due to individual treatment or combination treatment regimen
Progression-Free Survival (PFS) at 6 months | 6 months
  PFS at 6 months is defined as the percentage of participants who have neither progressed nor died within 6 months after the first dose of individual treatment or combination treatment regimen. PFS at 6 months will be assessed by (modified) Response assessment in neuro-oncology criteria (RANO) and estimated using Kaplan Meier method.
Progression-Free Survival (PFS) | Up to 5 years.
  PFS period is defined as the number of days from start of individual treatment or combination treatment regimen to disease progression or death. The PFS days of patient groups will be estimated using Kaplan-Meier method to show median progression-free period (days when 50% patients remain progression-free).
Time to Treatment Failure (TTF) | Up to 5 years
  Time to treatment failure is defined as the time from start of treatment to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death.
Overall survival (OS) | Up to 5 years
  Overall survival is defined as the length of time from start of individual treatment or combination treatment regimen until date of death. For the participants who were alive at the end of study or lost to follow-up, overall survival will be censored on the last date when participants were known to be alive. OS will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Clarke, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with study collaborators during the course of the study.

REFERENCES:
- [Background] Chen J, Oberheim Bush NA, Grabowsky JA, Kline C, Kroetz DL, Taylor JW, Villanueva-Meyer J, Molinaro AM, de Groot JF, Butowski NA, Tedesco M, Rabbitt J, Phillips JJ, Hervey-Jumper S, Aghi MK, Berger MS, Chang EF, Chang SM, Solomon DA, Clarke JL. A genomically-tailored multi-agent precision medicine clinical trial for adults with recurrent glioblastoma. Clin Cancer Res. 2026 Feb 6. doi: 10.1158/1078-0432.CCR-25-4080. Online ahead of print. PMID 41649856